CLINICAL TRIAL: NCT01312766
Title: Safety and Efficacy Study Comparing a New hMG Formulation (hMG-IBSA) to a Reference Product (Menopur®) in Patients Undergoing Ovarian Stimulation for in Vitro Fertilisation (IVF)
Brief Title: Safety and Efficacy Study in in Vitro Fertilisation (IVF) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10EU/hMG02; 2010-021021-13 (EudraCT Number)
Record Dates: First submitted 2011-03-07; First posted 2011-03-11 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Menotropins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- hMG-IBSA (Experimental): New hMG preparation.
  Interventions: Drug: Menotropins
- Menopur (Active Comparator)
  Interventions: Drug: Menotropins

INTERVENTIONS:
Drug: Menotropins — Daily administration, SC, starting dose 150 IU or 225 IU depending on patient age.
  Arms: hMG-IBSA
Drug: Menotropins — Daily administration, SC, starting dose 150 IU or 225 IU depending on patient age.
  Arms: Menopur

SUMMARY:
The purpose of the non-inferiority study is to evaluate the clinical efficacy and the safety of two different subcutaneous hMG preparations when administered to patients undergoing controlled ovarian stimulation for IVF.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing ovarian stimulation for IVF with the following characteristics:

  * Able and willing to sign the Patient Consent Form and adhere to the study visitation schedule
  * >18 and <40 years old
  * BMI between 18 and 30 kg/m2
  * less than 3 previously completed IVF cycles (i.e. completed cycle = egg recovery)
  * basal FSH <10 IU/L and E2 <80 pg/ml (~290 pmol/l)
  * Within 12 months of the beginning of the study, uterine cavity consistent with expected normal function as assessed through transvaginal ultrasound, hysterosalpingogram, sonohysterogram or hysteroscopic examination
  * Successful down-regulation performed with a standard GnRH-Agonist long protocol (Criteria for successful down-regulation: endometrial thickness < 7mm or serum E2 level <50 pg/ml (~185 pmol/l).

Exclusion Criteria:

* age <18 and >40 years
* primary ovarian failure or women known as poor responders (i.e. requiring more than 225 IU of hMG as a starting dose in previous treatment cycles or having less than 3 oocytes retrieved, or with a pre-ovulatory E2 serum concentration <500pg/ml (~1800 pmol/l))
* PCOS
* one or both ovaries inaccessible for oocyte retrieval
* ovarian cysts >10 mm
* hydrosalpinx that have not been surgically removed or ligated;
* stage 3 or 4 endometriosis
* oocyte donation
* implantation of previously frozen embryos
* patients affected by pathologies associated with any contraindication of being pregnant
* hypersensitivity to the study medication
* abnormal bleeding of undetermined origin
* uncontrolled thyroid or adrenal dysfunction
* neoplasias
* severe impairment of renal and/or hepatic function
* use of concomitant medications that might interfere with study evaluations (e.g. non-study hormonal medications, prostaglandin inhibitors, psychotropic agents)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2011-02; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique De Ziegler, MD, Prof, Principal Investigator — Hopital Cochin
Locations (6):
- Denmark (2):
  - Fertility clinic at Hvidovre Hospital, Hvidovre, Copenhagen
  - Odense Universitetshospital, Odense, Odensee C
- Groupe Hospitalier Cochin - Saint Vincent de Paul, Paris, France
- First Dept. Obstetric and Gynaecology, Semmelweiss University, Budapest, Hungary
- Universitätsspital Basel, Basel, Canton of Basel-City, Switzerland
- Midland Fertility Services, Aldridge, West Midlands, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | hMG-IBSA | Menopur
Started | 135 | 135
Completed | 129 | 130
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | hMG-IBSA | Menopur | Total
Number analyzed (Participants) | 135 | 135 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (4.0) | 33.0 (4.1) | 33.1 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 135 | 270
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 126 | 126 | 252
  Asian | 8 | 6 | 14
  Black | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Oocytes Retrieved
Time Frame: up to 24 days after treatment start
Measure: Mean (Standard Deviation); unit: number of oocytes
Arm/Group | hMG-IBSA | Menopur
Number analyzed (Participants) | 135 | 135
number of oocytes | 11.6 (6.6) | 9.7 (5.9)
Statistical Analysis 1: Comparison: hMG-IBSA vs Menopur; Test type: Non-Inferiority or Equivalence — The one-way Analysis of Variance with Least-Squares means was performed to calculate the 95% Confidence Interval of the difference between the two treatments. If the lower bound of the 95% Confidence Interval of the difference between means (hMG-IBSA minus Menopur®) was greater than -2.1, then hMG-IBSA would be considered to be not-inferior to the comparator; p = 0.012, ANOVA; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [0.43 to 3.43]

2. Secondary Outcome: Mean hMG Dose (Total);
Time Frame: up to 22 days after treatment start
Measure: Mean (Standard Deviation); unit: Internationa Units (IU)
Arm/Group | hMG-IBSA | Menopur
Number analyzed (Participants) | 135 | 135
Internationa Units (IU) | 2171.4 (980) | 2303.6 (906)
Statistical Analysis 1: Comparison: hMG-IBSA vs Menopur; Test type: Superiority or Other; p = 0.25, ANOVA

3. Secondary Outcome: Embryo Quality (Percentage of Patients With at Least One Top Quality Embryo)
Description: Assessed by counting the total number of embryos obtained, the number of embryos transferred, frozen and discarded.
Time Frame: up to 28 days after treatment start
Population: The population analysed corresponds to the patients who had at least one embryo to be analysed (i.e 120 participants in the hMG-IBSA group and 123 in the Menopur group). Of this, 119 in the hMG-IBSA group and 121 in the Menopur group underwent embryo transfer.
Measure: Number; unit: percentage of participants
Arm/Group | hMG-IBSA | Menopur
Number analyzed (Participants) | 120 | 123
percentage of participants | 63.3 (1.74) | 63.3 (1.65)

4. Secondary Outcome: Positive b-hCG Test
Time Frame: up to 5 weeks after treatment start
Measure: Number; unit: percentage of participants
Arm/Group | hMG-IBSA | Menopur
Number analyzed (Participants) | 135 | 135
percentage of participants | 43.7 | 45.2
Statistical Analysis 1: Comparison: hMG-IBSA vs Menopur; Test type: Superiority or Other; p = 0.90, Fisher Exact

5. Secondary Outcome: Controlled Ovarian Stimulation Duration (Days)
Time Frame: up to 23 days after treatment start
Measure: Mean (Standard Deviation); unit: days
Arm/Group | hMG-IBSA | Menopur
Number analyzed (Participants) | 135 | 135
days | 10.2 (1.3) | 10.6 (1.5)
Statistical Analysis 1: Comparison: hMG-IBSA vs Menopur; Test type: Superiority or Other; p = 0.02, ANOVA

6. Secondary Outcome: 17-β Estradiol (E2) Serum Concentration on the Monitoring Day Before hCG Injection;
Time Frame: up to 23 days after treatment start
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | hMG-IBSA | Menopur
Number analyzed (Participants) | 135 | 135
pg/ml | 2613.8 (1531.6) | 2364.0 (1441.6)

7. Secondary Outcome: Implantation Rate
Description: defined as the mean of the total number of implanted embryos (presence of gestational sac assessed by ultrasound) divided by the total number of transferred embryos x 100;
Time Frame: 10-11 weeks after embryo transfer
Measure: Mean (Standard Deviation); unit: percentage of embryos transferred
Arm/Group | hMG-IBSA | Menopur
Number analyzed (Participants) | 135 | 135
percentage of embryos transferred | 29.1 (41.0) | 28.2 (36.9)

8. Secondary Outcome: Clinical Pregnancy Rate,
Description: defined as a pregnancy showing ultrasound embryonic heart activity at 10 - 11 weeks after embryo transfer;
Time Frame: 10 - 11 weeks after embryo transfer
Measure: Number; unit: percentage of participants
Arm/Group | hMG-IBSA | Menopur
Number analyzed (Participants) | 135 | 135
percentage of participants | 33.3 | 37.1
Statistical Analysis 1: Comparison: hMG-IBSA vs Menopur; Test type: Superiority or Other; p = 0.61, Fisher Exact

9. Secondary Outcome: Number of Mature (Grade III Metaphase II) Oocytes Retrieved.
Time Frame: at the end of the stimulation.
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | hMG-IBSA | Menopur
Number analyzed (Participants) | 135 | 135
oocytes | 10.3 (6.0) | 8.2 (5.1)
Statistical Analysis 1: Comparison: hMG-IBSA vs Menopur; Test type: Superiority or Other; p = 0.002, ANOVA

10. Secondary Outcome: Ratio Mature/Total Number of Oocytes Retrieved.
Description: Percentage of retrieved oocytes considered to be mature.
Time Frame: at the end of the stimulation.
Measure: Number; unit: percentage of total oocytes retrieved
Arm/Group | hMG-IBSA | Menopur
Number analyzed (Participants) | 135 | 135
percentage of total oocytes retrieved | 85 | 81
Statistical Analysis 1: Comparison: hMG-IBSA vs Menopur; Test type: Superiority or Other; p = 0.004, ANOVA

11. Secondary Outcome: Total Number of Inseminated Oocytes (IVF and ICSI)
Description: number of oocytes that were inseminated via IVF or injected via ICSI technique.
Time Frame: on the day of oocyte retrieval
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | hMG-IBSA | Menopur
Number analyzed (Participants) | 135 | 135
oocytes | 10.8 (5.9) | 8.4 (5.0)
Statistical Analysis 1: Comparison: hMG-IBSA vs Menopur; Test type: Superiority or Other; p < 0.001, ANOVA

12. Secondary Outcome: Number of Cleaved Embryos
Time Frame: two days after insemination
Measure: Mean (Standard Deviation); unit: embryos
Arm/Group | hMG-IBSA | Menopur
Number analyzed (Participants) | 135 | 135
embryos | 5.8 (3.8) | 4.8 (3.7)
Statistical Analysis 1: Comparison: hMG-IBSA vs Menopur; Test type: Superiority or Other; p = 0.04, ANOVA

13. Secondary Outcome: Live Birth Rate
Time Frame: 9 months after treatment
Measure: Number; unit: percentage of participants
Arm/Group | hMG-IBSA | Menopur
Number analyzed (Participants) | 135 | 135
percentage of participants | 32.6 | 36.3
Statistical Analysis 1: Comparison: hMG-IBSA vs Menopur; Test type: Superiority or Other; p = 0.61, Fisher Exact

ADVERSE EVENTS:
Arm/Group | hMG-IBSA | Menopur
Serious Adverse Events (participants affected / at risk) | 5/135 | 8/135
Other Adverse Events (participants affected / at risk) | 46/135 | 42/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hMG-IBSA (N=135) | Menopur (N=135)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
peritoneal heamorrage (Gastrointestinal disorders) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headacje (Nervous system disorders) | 1 (1) | 0 (0)
Abortion Incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion Missed (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OHSS (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Ovarina torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hMG-IBSA (N=135) | Menopur (N=135)
Abdominal distension (Gastrointestinal disorders) | 18 (23) | 14 (18)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 6 (9)
fatigue (General disorders) | 9 (10) | 8 (9)
Headache (Nervous system disorders) | 21 (33) | 20 (32)
Hot flushes (Vascular disorders) | 11 (13) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No